CLINICAL TRIAL: NCT06508463
Title: Phase I Trial of Systemic Administration of Vesicular Stomatitis Virus Genetically Engineered to Express NIS and Human Interferon, in Patients With Relapsed or Refractory Multiple Myeloma, Acute Myeloid Leukemia, Lymphomas, or Histiocytic/Dendritic Cell Neoplasms
Brief Title: Intravenous Vesicular Stomatitis Virus in Patients With Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1684 Arm E; R01CA262613 (NIH); P50CA186781 (NIH); NCI-2017-00049 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1684 (Other: Mayo Clinic); 16-005474 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Peripheral T Cell Lymphoma; Relapsed Peripheral T-Cell Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Anaplastic Large Cell Lymphoma; Mycosis Fungoides; Relapsed Anaplastic Large Cell Lymphoma; Relapsed Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; sodium-iodide symporter; X-Rays; Photons; cemiplimab; Immunoglobulin G; Disulfides; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E (VSV-IFNβ-NIS, ipilimumab, cemiplimab) - Peripheral T-cell lymphoma (PTCL) only (Experimental): PTCL patients receive VSV-IFNβ-NIS IV over 30 minutes on day 1, ipilimumab IV over 30 minutes on day -3 and cemiplimab IV over 30 minutes on day -3 in the absence of disease progression or unacceptable toxicity. Patients undergo SPECT, CT scan, PET scan throughout the study. Patients may undergo tumor biopsy, bone marrow biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Biological: Cemiplimab; Biological: Ipilimumab
- Group E (VSV-IFNβ-NIS, ipilimumab, cemiplimab) - PTCL Expansion Cohort (Experimental): PTCL patients receive VSV-IFNβ-NIS IV over 30 minutes on day 1, ipilimumab IV over 30 minutes on day -3 and cemiplimab IV over 30 minutes on day -3 in the absence of disease progression or unacceptable toxicity. Patients undergo SPECT, CT scan, PET scan throughout the study. Patients may undergo tumor biopsy, bone marrow biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Biological: Cemiplimab; Biological: Ipilimumab

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo SPECT/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter — Given IV
  Other Names: Oncolytic VSV-hIFNbeta-NIS; Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Voyager-V1; VSV-expressing hIFNb and NIS; VSV-hIFNb-NIS; VSV-hIFNbeta-NIS; VV1; VSV-hIFNβ-NIS
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Biological: Cemiplimab — Given IV
  Other Names: 1801342-60-8; Cemiplimab RWLC; Cemiplimab-rwlc; Immunoglobulin G4; Anti-(Human Programmed Cell Death Protein 1) (Human Monoclonal REGN2810 Heavy Chain); Disulfide with Human Monoclonal REGN2810 kappa-chain; Libtayo; REGN2810
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy

SUMMARY:
This phase I trial studies the best dose and side effects of recombinant vesicular stomatitis virus (VSV) carrying the human (h) sodium iodide symporter (NIS) and Interferon (IFN) beta (β) genes (VSV-hIFNβ-NIS) in combination with ipilimumab and cemiplimab in patients with T-cell lymphoma. A virus, called VSV-hIFNβ-NIS, which has been changed in a certain way, may be able to kill cancer cells without damaging normal cells. Immunotherapy with ipilmumab and cemiplimab may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: To determine the maximum tolerated dose (MTD) of VSV-hIFNβ-NIS in combination with ipilimumab and cemiplimab in patients with T-cell lymphoma [Group E].

Patients undergo computed tomography (CT) scan, position emission tomography (PET) scan throughout the study. Patients may undergo tumor biopsy, bone marrow biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 28 days, and then every 3 months for up to 1 year or until progressive disease, then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Relapsed or refractory:

  * Group E only: Relapsed peripheral T-cell lymphoma (PTCL) of the following histologies: peripheral T-cell lymphoma-NOS (PTCL-NOS); anaplastic large cell (ALCL), and mycosis fungoides (MF)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2 times upper limit of normal (ULN) (obtained =< 15 days prior to registration)
* Creatinine =< 2.0 mg/dL (obtained =< 15 days prior to registration)
* Direct bilirubin =< 1.5 x ULN (obtained =< 15 days prior to registration)
* International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (obtained =< 15 days prior to registration)
* If baseline liver disease, Child Pugh score not exceeding class A (obtained =< 15 days prior to registration)
* Negative pregnancy test for persons of child-bearing potential (obtained =< 15 days prior to registration)
* FOR T-Cell Lymphoma (TCL)/B-Cell Lymphoma (BCL) ONLY: Absolute Neutrophil Count (ANC) >= 1,000/microliter (μL) (obtained =< 14 days prior to registration)
* FOR TCL/BCL ONLY: Platelets >= 100,000/μL (obtained =< 14 days prior to registration)
* FOR TCL/BCL ONLY: Hemoglobin >= 8.5 g/dl (obtained =< 14 days prior to registration)
* FOR TCL/BCL ONLY: Measurable disease by CT or magnetic resonance imaging (MRI): must have at least one lesion that has a single diameter of > 2 cm or tumor cells in the blood > 5 x 10^9/L; NOTE: skin lesions can be used if the area is > 2 cm in at least one diameter and photographed with a ruler and the images are available in the medical record
* Absence of active central nervous system (CNS) involvement; NOTE: pre-enrollment lumbar puncture not mandatory
* Ability to provide written informed consent
* Willingness to return to Mayo Clinic for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Willing to provide mandatory biological specimens for research purposes

Exclusion Criteria:

* Availability of and patient acceptance of curative therapy
* Uncontrolled infection
* Active tuberculosis or hepatitis, or chronic hepatitis
* Any of the following prior therapies:

  * Chemotherapy (IMIDs, alkylating agents, proteosome inhibitors) =< 2 weeks prior to registration
  * Immunotherapy (monoclonal antibodies) =< 4 weeks prior to registration
  * Experimental agent in case of Acute Myeloid Leukemia (AML) or TCL within 4 half-lives of the last dose of the agent
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias [atrial fibrillation or supraventricular tachycardia (SVT)]
* Active CNS disorder or seizure disorder or known CNS disease or neurologic symptomatology; in case of AML active CNS involvement as detected by lumbar puncture or neuro-imaging (only to be done if clinically indicated)
* Human immunodeficiency virus (HIV) positive test result or other immunodeficiency or immunosuppression
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (used for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation);

  * NOTE: in TCL, patients may use topical emollients or corticosteroids, acetic acid soaks, etc. to control pruritis and prevent infection; no topical chemotherapy is allowed (no topical nitrogen mustard)
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women or women of reproductive ability who are unwilling to use effective contraception
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP E (COMBINATION WITH IPILIMUMAB AND CEMIPLIMAB) ONLY:

  * Diagnosis of AML
  * Diagnosis of Angioimmunoblastic T-cell Lymphoma (AITL)
  * Hypersensitivity to ipilimumab or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events of grade 3 or higher | Up to 2 years
  Assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Clinical response | Up to 2 years
  Response to treatment will be recorded as stringent Complete Response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), Minimal Response (MR), stable disease (SD), and progressive disease (PD).
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from study enrollment to disease progression or death due to any cause.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from study enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Whye Peng, PhD, Principal Investigator — Mayo Clinic in Rochester; Nora Bennani, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cook J, Peng KW, Witzig TE, Broski SM, Villasboas JC, Paludo J, Patnaik M, Rajkumar V, Dispenzieri A, Leung N, Buadi F, Bennani N, Ansell SM, Zhang L, Packiriswamy N, Balakrishnan B, Brunton B, Giers M, Ginos B, Dueck AC, Geyer S, Gertz MA, Warsame R, Go RS, Hayman SR, Dingli D, Kumar S, Bergsagel L, Munoz JL, Gonsalves W, Kourelis T, Muchtar E, Kapoor P, Kyle RA, Lin Y, Siddiqui M, Fonder A, Hobbs M, Hwa L, Naik S, Russell SJ, Lacy MQ. Clinical activity of single-dose systemic oncolytic VSV virotherapy in patients with relapsed refractory T-cell lymphoma. Blood Adv. 2022 Jun 14;6(11):3268-3279. doi: 10.1182/bloodadvances.2021006631. PMID 35175355
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials